CLINICAL TRIAL: NCT06015750
Title: An Interventional, Prospective Open-Label Study of Immunosuppressive Therapies to Mitigate Immune-Mediated Loss of Therapeutic Response to Asfotase Alfa (STRENSIQ®) for Hypophosphatasia (RESTORE)
Brief Title: Mitigate Immune-Mediated Loss of Therapeutic Response to Asfotase Alfa (STRENSIQ®) for Hypophosphatasia
Acronym: RESTORE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision following FDA release from the PMR.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8400C00001; AA-HPP-407 (Other: Alexion); 2022-502793-17 (EudraCT Number)
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Asfotase alfa; Strensiq
MeSH Terms: conditions — Hypophosphatasia | interventions — Methotrexate; Rituximab; Bortezomib; Immunoglobulins, Intravenous; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pediatric participants with HPP (Experimental): Pediatric participants who have been receiving asfotase alfa treatment for their HPP, and who demonstrate immune-mediated LoE.
  Interventions: Drug: methotrexate; Drug: rituximab; Drug: bortezomib; Drug: IVIg; Drug: Folic Acid

INTERVENTIONS:
Drug: methotrexate — Methotrexate will be administered SC or orally weekly for 104 weeks.
Drug: rituximab — Rituximab will be administered intravenously (IV) continuously weekly, for up to 74 weeks.
Drug: bortezomib — Bortezomib will be administered via IV bolus or SC, as needed.
Drug: IVIg — IVIg will be administered via IV monthly through initial 74 weeks.
Drug: Folic Acid — Folic acid will be given orally as long as methotrexate is being dosed.

SUMMARY:
The primary objective of this study is to evaluate the effect of immunosuppressive therapy (IST) in participants treated with asfotase alfa who demonstrate immune-mediated loss of effectiveness (LoE).

DETAILED DESCRIPTION:
The administration of biological drugs to patients, especially for chronic conditions, carries a risk of eliciting anti-drug antibodies. Neutralizing antibodies can neutralize the clinical benefit of the agent. In postmarketing safety surveillance, some patients treated with asfotase alfa demonstrated an initial response, but subsequently recurrence and progression of disease. Consequently, the FDA requested a study to assess a potential serious risk of immune-mediated loss of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Reoccurrence or worsening of rickets for at least the past 3 months in participants who showed an initial efficacy response to asfotase alfa after at least 6 months of continuous treatment and currently receiving asfotase alfa. RSS will be used to determine severity at Baseline.
* Presence of ADAs, with or without NAbs, irrespective of their titers.
* Confirmation by the TMB that both the clinical evidence and immunogenicity-mediated association noted above are present.
* Female participants of childbearing potential and male participants with partners of childbearing potential must follow protocol-specified contraception guidance as described in Section 10.5.
* Participant, or participant's legal guardian, is capable of signing informed consent or assent as described in Section 10.1.3, which includes compliance with the requirements and restrictions listed in the informed consent or assent form and in this protocol.

Exclusion Criteria:

* Known history of human immunodeficiency virus (HIV) infection (evidenced by HIV type 1 or type 2 [HIV 1, HIV 2] antibody) or hepatitis B or C viral infection.
* Known or suspected history of drug or alcohol abuse or dependence within 1 year prior to Screening.
* Inability of the participant, or the participant's legal guardian, to provide informed consent.
* Pregnant, breastfeeding, or intending to conceive during the course of the study.
* Inability to travel to the clinic for specified visits during the Treatment Period caused by disease per se or logistics (does not apply to external travel restrictions).
* The participant is at risk of reactivation or has an active significant viral infection such as hepatitis B, cytomegalovirus, herpes simplex, human polyomavirus (also known as John Cunningham [JC] virus), parvovirus, or Epstein Barr virus.
* The participant is at risk of reactivation of tuberculosis or has regular contact (eg, in the household) with individuals who are being actively treated for tuberculosis.
* The participant has had or is required to have any live vaccination within 1 month prior to enrollment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2026-07-29 (Estimated); Primary Completion 2030-03-13 (Estimated); Study Completion 2030-03-13 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Achieve Immunosuppressive Therapy (IST) Complete Response at Week 100 | Week 100

SECONDARY OUTCOMES:
Number Participants with Antidrug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) | Baseline Through Week 100
ADA and NAb Titer Levels | Baseline Through Week 100
Serum Concentration of Asofatase Alfa (Measured as Enzyme Activity) | Baseline Through Week 100
Plasma Concentration of Pyridoxal-5ˈ-Phosphate (PLP) | Baseline Through Week 100
Plasma Concentration of Inorganic Pyrophosphates (PPi) | Baseline Through Week 100
Number of Participants with Treatment-emergent Adverse Events and Treatment-emergent Serious Adverse Events | Baseline Through Week 104

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR